CLINICAL TRIAL: NCT03694002
Title: A Randomized Phase II Trial of Carboplatin-Paclitaxel With or Without Ramucirumab in Patients With Unresectable Locally Advanced, Recurrent, or Metastatic Thymic Carcinoma
Brief Title: Carboplatin and Paclitaxel With or Without Ramucirumab in Treating Patients With Locally Advanced, Recurrent, or Metastatic Thymic Cancer That Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S1701; NCI-2017-02254 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S1701; S1701 (Other: SWOG); S1701 (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2018-10-01; First posted 2018-10-03 (Actual); Results first posted 2025-10-30 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Locally Advanced Thymic Carcinoma; Metastatic Thymic Carcinoma; Recurrent Thymic Carcinoma; Unresectable Thymic Carcinoma
MeSH Terms: conditions — Thymoma | interventions — Carboplatin; Paclitaxel; Taxes; Ramucirumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (ramucirumab, carboplatin, paclitaxel) (Experimental): Patients receive ramucirumab IV over 60 minutes, carboplatin IV, and paclitaxel IV on day 1. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients who have not progressed may continue to receive ramucirumab for up to 1 year.
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Biological: Ramucirumab
- Arm B (carboplatin, paclitaxel) (Active Comparator): Patients receive carboplatin IV and paclitaxel IV on day 1. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Biological: Ramucirumab — Given IV
  Other Names: Anti-VEGFR-2 Fully Human Monoclonal Antibody IMC-1121B; Cyramza; IMC-1121B; LY3009806; Monoclonal Antibody HGS-ETR2
  Arms: Arm A (ramucirumab, carboplatin, paclitaxel)

SUMMARY:
This randomized phase II trial studies how well carboplatin and paclitaxel with or without ramucirumab work in treating patients with thymic cancer that has spread to other places in the body, has come back, or cannot be removed by surgery. Drugs used in chemotherapy, such as carboplatin and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Monoclonal antibodies, such as ramucirumab, may interfere with the ability of tumor cells to grow and spread. It is not yet known if giving carboplatin and paclitaxel with or without ramucirumab will work better in treating patients with thymic cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare progression-free survival between patients with incurable unresectable locally advanced, or recurrent, or metastatic thymic carcinoma randomized to carboplatin-paclitaxel with or without ramucirumab.

SECONDARY OBJECTIVES:

I. To evaluate the frequency and severity of toxicity of carboplatin-paclitaxel with or without ramucirumab in this patient population.

II. To compare the response rate (complete response, partial response, confirmed and unconfirmed) between treatment arms.

III. To compare disease control rate (complete response, partial response, confirmed or unconfirmed, stable disease) between treatment arms.

IV. To compare overall survival between treatment arms.

ADDITIONAL OBJECTIVE:

I. To bank specimens for future research.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive ramucirumab intravenously (IV) over 60 minutes, carboplatin IV, and paclitaxel IV on day 1. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients who have not progressed may continue to receive ramucirumab for up to 1 year.

ARM B: Patients receive carboplatin IV and paclitaxel IV on day 1. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 1 year, and then every 6 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed thymic carcinoma; thymic carcinoma may be defined as "thymic epithelial malignancy, consistent with thymic carcinoma", or "World Health Organization (WHO) type C thymic epithelial tumor", or "thymic epithelial malignancy" with radiographic imaging consistent with thymic carcinoma
* Patients must have unresectable thymic carcinoma, that is either locally advanced, recurrent, or metastatic
* Patients must not be candidates for localized surgery
* Patients must have measurable disease documented by computed tomography (CT) or magnetic resonance imaging (MRI) within 28 calendar days prior to randomization; the CT from a combined positron emission tomography (PET)/CT may be used only if it is of diagnostic quality; non-measurable disease must be assessed within 42 calendar days prior to randomization; all known sites of disease must be assessed and documented on the baseline tumor assessment form (Response Evaluation Criteria in Solid Tumors [RECIST] 1.1)
* Patients must have a Zubrod performance status of 0 to 2
* Patients must not have undergone major surgery within 28 calendar days prior to randomization, or minor surgery/subcutaneous venous access device placement within 7 calendar days prior to randomization; the patient must not have elective or planned major surgery to be performed during the course of the clinical trial
* Patients must not have had prior systemic anti-cancer therapy for locally advanced or metastatic unresectable thymic carcinoma
* If patients have recurrent unresectable thymic carcinoma, patients may have had prior neoadjuvant or adjuvant chemotherapy if treatment concluded >= 6 months prior to randomization
* Patients must have a CT or MRI scan of the brain to evaluate for central nervous system (CNS) disease within 42 calendar days prior to registration; patient must not have brain metastases unless: (1) metastases have been treated and have remained controlled for at least two weeks following treatment, AND (2) patient has no residual neurological dysfunction off corticosteroids for at least 1 day
* Patients must not be candidates for radiation therapy with curative intent; prior palliative radiation therapy is allowed as long as a period of 7 days has passed since the last dose was received and the patient has recovered from any associated toxicity at the time of randomization
* Absolute neutrophil count (ANC) >= 1500/mcL documented within 28 calendar days prior to randomization
* Hemoglobin >= 9 g/dL (5.58 mmol/L) documented within 28 calendar days prior to randomization
* Platelets >= 100,000/mcL documented within 28 calendar days prior to randomization
* International normalized ratio (INR) =< 1.5 documented within 28 calendar days prior to randomization
* Partial thromboplastin time (PTT) =< 5 seconds above the institutional upper limit of normal (IULN) (unless receiving anticoagulation therapy) documented within 28 calendar days prior to randomization
* Patients receiving warfarin must be switched to low molecular weight heparin and have achieved stable coagulation profile 14 days prior to randomization
* Patients must not have experienced any grade 3 or above gastrointestinal (GI) bleeding within 84 calendar days prior to randomization
* Patients must not have a history of deep vein thrombosis (DVT), pulmonary embolism (PE), or any other significant thromboembolism (venous port or catheter thrombosis or superficial venous thrombosis are not considered "significant") during the 84 calendar days prior to randomization
* Total bilirubin =< 1.5 x the institutional upper limit normal (IULN) documented within 28 calendar days prior to randomization
* Aspartate aminotransferase (aspartate transaminase [AST]) and alanine aminotransferase (alanine transaminase [ALT]) =< 3.0 x IULN; for patients with liver metastases, total bilirubin and AST or ALT must be =< 5.0 x IULN documented within 28 calendar days prior to randomization
* Patients must not have any of following:

  * Cirrhosis at a level of Child-Pugh B (or worse)
  * Cirrhosis (any degree) and a history of hepatic encephalopathy; or
  * Clinically meaningful ascites resulting from cirrhosis; clinically meaningful ascites is defined as ascites from cirrhosis requiring diuretics or paracentesis
* Serum creatinine =< 1.5 x IULN, or creatinine clearance (measured via 24-hour urine collection) >= 40 mL/minute (that is, if serum creatinine is > 1.5 x ULN, a 24-hour urine collection to calculate creatinine clearance must be performed) documented within 28 calendar days prior to randomization
* Patient urinary protein must be =< 1+ on dipstick or routine urinalysis (UA); if urine dipstick or routine analysis is >= 2+, a 24-hour urine collection for protein must demonstrate < 1000 mg of protein in 24 hours); these tests must be documented within 28 calendar days prior to randomization
* Patients must not have experienced any arterial thromboembolic events, including but not limited to myocardial infarction, transient ischemic attack, cerebrovascular accident, or unstable angina, within 6 months prior to randomization
* Patients must not have a history of uncontrolled or poorly-controlled hypertension (defined as > 160 mmHg systolic or > 100 mmHg diastolic for > 4 weeks) despite standard medical management
* Patients must not be pregnant or nursing; women/men of reproductive potential must have agreed to use an effective contraceptive method (hormonal or barrier method of birth control; abstinence) prior to randomization, during the study participation and for 4 months after the last dose of protocol treatment; a woman is considered to be of "reproductive potential" if she has had menses at any time in the preceding 12 consecutive months; in addition to routine contraceptive methods, "effective contraception" also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy or bilateral tubal ligation; however, if at any point a previously celibate patient chooses to become heterosexually active during the time period for use of contraceptive measures outlined in the protocol, he/she is responsible for beginning contraceptive measures
* Patients must not have experienced hemoptysis (defined as bright red blood or >= 1/2 teaspoon) within 2 months prior to randomization or with radiographic evidence of intratumor cavitation or has radiologically documented evidence of major blood vessel invasion or encasement by cancer
* Patients must not have a prior history of gastrointestinal perforation/fistula (within 6 months of randomization) or risk factors for perforation
* Patients must not have a serious or nonhealing wound, ulcer, or bone fracture within 28 calendar days prior to randomization
* Patients must not be receiving chronic antiplatelet therapy, including aspirin, nonsteroidal anti-inflammatory drugs (NSAIDs, including ibuprofen, naproxen, and others), dipyridamole or clopidogrel, or similar agents within 7 days prior to randomization; once-daily aspirin use (maximum dose 325 mg/day) is permitted
* Patients must be offered the opportunity to participate in banking of specimens for future research
* Patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* As a part of the Oncology Patient Enrollment Network (OPEN) registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne S Tsao, Principal Investigator — SWOG Cancer Research Network
Locations (254):
- United States (254):
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Kingman Regional Medical Center, Kingman, Arizona
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - Mission Hope Medical Oncology - Arroyo Grande, Arroyo Grande, California
  - PCR Oncology, Arroyo Grande, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - City of Hope Antelope Valley, Lancaster, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - City of Hope Mission Hills, Mission Hills, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Mission Hope Medical Oncology - Santa Maria, Santa Maria, California
  - City of Hope South Pasadena, South Pasadena, California
  - City of Hope West Covina, West Covina, California
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Southwest Oncology PC, Durango, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Moffitt Cancer Center-International Plaza, Tampa, Florida
  - Moffitt Cancer Center - McKinley Campus, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Medical Center, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Medical Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Cancer Center, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Northwestern University, Chicago, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - Jewish Hospital Medical Center Northeast, Louisville, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Allegiance Health, Jackson, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - Henry Ford Macomb Health Center - Shelby Township, Shelby, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Hospital, Missoula, Montana
  - CHI Health Saint Francis, Grand Island, Nebraska
  - Heartland Hematology and Oncology, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hematology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Horizon Ridge, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - 21st Century Oncology-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Las Vegas Urology - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pebble, Henderson, Nevada
  - Urology Specialists of Nevada - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pecos, Las Vegas, Nevada
  - Desert West Surgery, Las Vegas, Nevada
  - OptumCare Cancer Care at Oakey, Las Vegas, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Hope Cancer Care of Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - Urology Specialists of Nevada - Central, Las Vegas, Nevada
  - 21st Century Oncology, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Las Vegas Prostate Cancer Center, Las Vegas, Nevada
  - Las Vegas Urology - Sunset, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - 21st Century Oncology-Vegas Tenaya, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Las Vegas Urology - Cathedral Rock, Las Vegas, Nevada
  - Las Vegas Urology - Smoke Ranch, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Urology Specialists of Nevada - Northwest, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Town Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - 21st Century Oncology-Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Urology Specialists of Nevada - Southwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - University Cancer Center, Las Vegas, Nevada
  - Hope Cancer Care of Nevada-Pahrump, Pahrump, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - NYP/Weill Cornell Medical Center, New York, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Saint Alphonsus Medical Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Medical Center-Ontario, Ontario, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Prisma Health Cancer Institute - Spartanburg, Spartanburg, South Carolina
  - Memorial Hospital, Chattanooga, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - Overlake Medical Center, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Harrison Medical Center, Bremerton, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Valley Medical Center, Renton, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Marshfield Clinic - Ladysmith Center, Ladysmith, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Marshfield Clinic Stevens Point Center, Stevens Point, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 21 participant enrolled, 20 of which were eligible. 3 participants withdrew consent before treatment start.
Groups:
- Experimental: Arm A (Ramucirumab, Carboplatin, Paclitaxel): Patients receive ramucirumab IV over 60 minutes, carboplatin IV, and paclitaxel IV on day 1. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients who have not progressed may continue to receive ramucirumab for up to 1 year.
- Active Comparator: Arm B (Carboplatin, Paclitaxel): Patients receive carboplatin IV and paclitaxel IV on day 1. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Experimental: Arm A (Ramucirumab, Carboplatin, Paclitaxel) | Active Comparator: Arm B (Carboplatin, Paclitaxel)
Started | 8 | 13
Completed | 1 | 7
Not Completed | 7 | 6
Not completed — Progression | 4 | 2
Not completed — Adverse Event | 2 | 0
Not completed — Other not protocol specified | 1 | 0
Not completed — Ineligible | 0 | 1
Not completed — Withdrew consent before starting treatment | 0 | 3

BASELINE CHARACTERISTICS:
Population: All eligible participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental: Arm A (Ramucirumab, Carboplatin, Paclitaxel) | Active Comparator: Arm B (Carboplatin, Paclitaxel) | Total
Number analyzed (Participants) | 8 | 12 | 20
Age, Continuous [Median (Full Range); unit: Years] | 68.2 [31.7 to 72.3] | 65.7 [28.4 to 73.5] | 66.8 [28.4 to 73.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 7 | 8 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 6 | 7 | 13
  Black | 0 | 2 | 2
  Asian | 0 | 2 | 2
  Unknown | 2 | 1 | 3
Hispanic [Count of Participants; unit: Participants]
  Yes | 3 | 1 | 4
  No | 5 | 10 | 15
  Unknown | 0 | 1 | 1
Performance Status [Count of Participants; unit: Participants] — Performance Status Scores:
  0 - Fully active, able to carry on all pre-disease performance without restriction.
  1 - Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework, office work.
  Participants
    0 | 5 | 8 | 13
    1 | 3 | 4 | 7
Pathologic cancer type [Count of Participants; unit: Participants]
  Thymic epithelial malignancy | 1 | 2 | 3
  Thymic carcinoma, not otherwise specified | 5 | 10 | 15
  Unknown | 2 | 0 | 2
Histologic subtype [Count of Participants; unit: Participants]
  Squamous cell | 6 | 10 | 16
  Lymphoepithelioma like | 0 | 1 | 1
  Undifferentiated | 2 | 1 | 3
Palliative radiation therapy [Count of Participants; unit: Participants]
  Yes | 0 | 1 | 1
  No | 8 | 11 | 19
Neoadjuvant chemotherapy [Count of Participants; unit: Participants]
  Yes | 1 | 0 | 1
  No | 7 | 12 | 19
Adjuvant chemotherapy [Count of Participants; unit: Participants]
  Yes | 1 | 1 | 2
  No | 7 | 11 | 18

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Compare progression-free survival between patients with incurable unresectable locally advanced, or recurrent, or metastatic thymic carcinoma randomized to carboplatin-paclitaxel with or without ramucirumab. Progression-free survival is defined as: From date of registration to date of first documentation of progression or symptomatic deterioration, or death due to any cause.
  Progression is defined as: 20% increase in the sum of appropriate diameters of target measurable lesions over smallest sum observed, as well as an absolute increase of at least 0.5 cm. Unequivocal progression of non-measurable disease in the opinion of the treating physician (an explanation must be provided). Appearance of any new lesion/site. Death due to disease without prior documentation of progression and without symptomatic deterioration
Time Frame: up to 2 years after registration
Population: All eligible participants who received at least one cycle of treatment.
Measure: Median (80% Confidence Interval); unit: Months
Arm/Group | Experimental: Arm A (Ramucirumab, Carboplatin, Paclitaxel) | Active Comparator: Arm B (Carboplatin, Paclitaxel)
Number analyzed (Participants) | 8 | 12
Months | 8 [7 to 11] | 7 [6 to 8]

2. Secondary Outcome: Frequency and Severity of Adverse Events
Description: Only adverse events that are possibly, probably or definitely related to study drug are reported.
Time Frame: Up to 2 years post randomization
Population: Participants who received any protocol treatment
Measure: Number; unit: Participants
Arm/Group | Experimental: Arm A (Ramucirumab, Carboplatin, Paclitaxel) | Active Comparator: Arm B (Carboplatin, Paclitaxel)
Number analyzed (Participants) | 8 | 9
Participants
  Anemia | 1 | 0
  Diarrhea | 1 | 0
  Dyspnea | 1 | 0
  Ejection fraction decreased | 1 | 0
  Fatigue | 1 | 0
  Lymphocyte count decreased | 1 | 0
  Neutrophil count decreased | 0 | 1
  Resp, thoracic and mediastinal disorders - Other | 1 | 0
  Thromboembolic event | 0 | 1
  White blood cell decreased | 1 | 1

3. Secondary Outcome: Response Rate
Description: To compare the response rate (complete response, partial response, confirmed and unconfirmed) between treatment arms in the subset of this patient population with measurable disease.
  Complete response - Complete disappearance of all target and non-target lesions (with the exception of lymph nodes mentioned below). No new lesions. No disease related symptoms. Any lymph nodes (whether target or non-target) must have reduction in short axis to < 1.0 cm.
  Partial response - Applies only to patients with at least 1 measurable lesion. Greater than or equal to 30% decrease under baseline of the sum of appropriate diameters of all targets measurable lesions. No unequivocal progression of non-measurable disease. No new lesions.
Time Frame: Up to 2 years after registration
Population: Participants who had measurable disease. 2 participants in the active comparator arm did not have measurable disease.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Arm A (Ramucirumab, Carboplatin, Paclitaxel) | Active Comparator: Arm B (Carboplatin, Paclitaxel)
Number analyzed (Participants) | 8 | 10
Participants
  Complete response | 0 | 0
  Partial repsonse | 7 | 4
  No response | 1 | 6

4. Secondary Outcome: Disease Control Rate
Description: To compare disease control rate (complete response, partial response, confirmed or unconfirmed, stable disease) between treatment arms in the subset of this patient population with measurable disease.
Time Frame: Up to 2 years after registration
Population: Participants with measurable disease and achieved a response. 2 participants in the active comparator arm had non-measurable disease. 6 participants in the active comparator arm had no response and 1 participants in the experimental arm had no response.
Measure: Median (Full Range); unit: months
Arm/Group | Experimental: Arm A (Ramucirumab, Carboplatin, Paclitaxel) | Active Comparator: Arm B (Carboplatin, Paclitaxel)
Number analyzed (Participants) | 7 | 4
months | 2.92 [1.4 to 3.23] | 1.67 [1.47 to 6.43]

5. Secondary Outcome: Overall Survival
Description: To compare overall survival between treatment arms. Overall survival is defined as time from date of registration to date of death due to any cause. Because of low accrual, and too few participant deaths, we do not plan to analyze or report with outcome.
Time Frame: Up to 2 years after registration
Population: Only one death has been reported - so this outcome can not be completed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Experimental: Arm A (Ramucirumab, Carboplatin, Paclitaxel) | Active Comparator: Arm B (Carboplatin, Paclitaxel)
Number analyzed (Participants) | 8 | 12
months | NA [NA to NA] — could not be calculated due to an insufficient number of events | NA [NA to NA] — could not be calculated due to an insufficient number of events

ADVERSE EVENTS:
Time Frame: Up to 2 years after randomization
Arm/Group | Experimental: Arm A (Ramucirumab, Carboplatin, Paclitaxel) | Active Comparator: Arm B (Carboplatin, Paclitaxel)
All-Cause Mortality (participants affected / at risk) | 1/8 | 2/9
Serious Adverse Events (participants affected / at risk) | 3/8 | 0/9
Other Adverse Events (participants affected / at risk) | 8/8 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: Arm A (Ramucirumab, Carboplatin, Paclitaxel) (N=8) | Active Comparator: Arm B (Carboplatin, Paclitaxel) (N=9)
Anal ulcer (Gastrointestinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: Arm A (Ramucirumab, Carboplatin, Paclitaxel) (N=8) | Active Comparator: Arm B (Carboplatin, Paclitaxel) (N=9)
Anemia (Blood and lymphatic system disorders) | 2 | 1
Cardiac disorders-Other (Cardiac disorders) | 1 | 1
Palpitations (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0
Blurred vision (Eye disorders) | 2 | 0
Dry eye (Eye disorders) | 1 | 0
Eye disorders-Other (Eye disorders) | 1 | 0
Floaters (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 0
Bloating (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 3 | 3
Diarrhea (Gastrointestinal disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 5 | 4
Vomiting (Gastrointestinal disorders) | 1 | 1
Chills (General disorders) | 0 | 1
Edema limbs (General disorders) | 1 | 0
Fatigue (General disorders) | 7 | 4
Fever (General disorders) | 0 | 2
General disorders and admin site conditions - Other (General disorders) | 2 | 0
Infusion related reaction (General disorders) | 1 | 0
Pain (General disorders) | 3 | 1
Infections and infestations-Other (Infections and infestations) | 2 | 1
Upper respiratory infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 1
Alanine aminotransferase increased (Investigations) | 1 | 1
Alkaline phosphatase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0
Ejection fraction decreased (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 1 | 2
Neutrophil count decreased (Investigations) | 2 | 1
Platelet count decreased (Investigations) | 1 | 0
Weight loss (Investigations) | 1 | 0
White blood cell decreased (Investigations) | 3 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Musculoskeletal and connective tiss disorder - Other (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1
Dizziness (Nervous system disorders) | 3 | 0
Dysgeusia (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 0
Nervous system disorders-Other (Nervous system disorders) | 0 | 1
Paresthesia (Nervous system disorders) | 3 | 1
Peripheral motor neuropathy (Nervous system disorders) | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 4
Sinus pain (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1
Hematuria (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 2 | 0
Renal and urinary disorders-Other (Renal and urinary disorders) | 1 | 0
Renal calculi (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Urinary tract pain (Renal and urinary disorders) | 1 | 0
Urinary urgency (Renal and urinary disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Resp, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 2
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 | 1
Hypertension (Vascular disorders) | 2 | 1
Thromboembolic event (Vascular disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-07-27): https://cdn.clinicaltrials.gov/large-docs/02/NCT03694002/Prot_SAP_000.pdf
  • Informed Consent Form (2022-07-27): https://cdn.clinicaltrials.gov/large-docs/02/NCT03694002/ICF_001.pdf